CLINICAL TRIAL: NCT03393611
Title: A Pilot Study of a Novel Sequential Treatment Utilizing CPX-351 as Salvage Chemotherapy Followed by Allogeneic Stem-Cell Transplantation (SCT) Utilizing a Haplo-cord Graft for Patients With Relapsed or Refractory Leukemia or Myelodysplastic Syndrome
Brief Title: CPX-351 Salvage Therapy Followed by Haplo-Cord Transplant for Relapsed/Refractory Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1107011830
Record Dates: First submitted 2017-12-07; First posted 2018-01-08 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Relapsed Adult Acute Myeloid; Myelodysplastic Syndromes, Previously Treated
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia | interventions — CPX-351; fludarabine; fludarabine phosphate; Melphalan; Antilymphocyte Serum; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPX-351 Salvage Therapy and Transplant (Experimental): Subjects will receive CPX-351 salvage chemotherapy on Day -21, -19, and -17 as a bridge to allogeneic stem cell transplantation using a Fludarabine/Melphalan/rATG conditioning regimen and a haplo-cord graft.
  Interventions: Drug: CPX-351; Drug: Fludarabine; Drug: Melphalan; Drug: Rabbit Anti-Human T-Lymphocyte Globulin; Biological: Haplo-Cord Stem Cell Transplantation

INTERVENTIONS:
Drug: CPX-351 — Salvage Chemotherapy: CPX-351 at 120 u/m2 on Days -21, -19, and -17
  Other Names: Cytarabine:Daunorubicin Liposome Injection
Drug: Fludarabine — Fludarabine 150 mg/m2 (30 mg/m2/day x 5 days, Day -7 to Day -3)
  Other Names: Fludara
Drug: Melphalan — Melphalan 140 mg/m2 (Day -2)
  Other Names: Alkeran
Drug: Rabbit Anti-Human T-Lymphocyte Globulin — Rabbit ATG (rATG)-thymoglobulin 4.5 mg/kg (1.5 mg/kg/day x 3 days)
  Other Names: Thymoglobulin
Biological: Haplo-Cord Stem Cell Transplantation — Allogeneic stem cell transplantation using a haploidentical donor and umbilical cord blood unit.

SUMMARY:
This pilot study is designed to evaluate outcomes with the combination of CPX-351 salvage therapy and haplo-cord graft stem cell transplantation for subjects with relapsed or refractory AML or myelodysplastic syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have refractory or relapsed Acute Myeloid Leukemia (AML) according to previously established criteria:

   1. Primary induction failure (PIF) after ≥ 2 cycles of chemotherapy
   2. First relapse
   3. Relapse refractory to salvage chemotherapy
   4. Second or subsequent relapse
2. Subjects with Myelodysplastic Syndrome (MDS):

   (a) Either Refractory Anemia with Excess Blasts I or Refractory Anemia with Excess Blasts II (RAEB I or RAEB II)
3. Karnofsky performance status ≥ 70
4. Willing to participate as a research subject and sign an informed consent form
5. Adequate physical function measured by:

   1. Cardiac: asymptomatic, or if symptomatic then Left Ventricular Ejection Fraction (LVEF) at rest must be ≥ 45% and must improve with exercise
   2. Hepatic: ≤3 x upper limit of normal (ULN) alanine aminotransferase (ALT) and ≤ 1.5 total serum bilirubin, unless liver is involved with the disease or there is congenital benign hyperbilirubinemia
   3. Renal: serum creatinine within normal range, or if serum creatinine is outside the normal range, then calculated creatinine clearance ≥ 60 ml/min
   4. Pulmonary: asymptomatic, or if symptomatic, diffusing capacity of the lungs for carbon monoxide (DLCO) ≥ 45% of predicted (corrected for hemoglobin)
6. If subject has prior malignancy, must be without any evidence of disease of that prior malignancy for at least 2 years (excludes skin cancers that may have been excised within that 2 year period).

Exclusion Criteria:

1. Serious active or uncontrolled infection or medical condition
2. Women who are pregnant or breast feeding. Women of childbearing age must use adequate contraception and have a negative pregnancy test.
3. Prior daunorubicin therapy with a cumulative dose of more than 368 mg/m2 or equivalent
4. Other systemic anticancer therapy or ongoing clinically relevant toxicities from such therapy (at discretion of the investigator)
5. History of and/or current evidence of myocardial impairment (e.g. cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, congestive heart failure), resulting in heart failure by New York Heart Association Class III or IV staging.
6. Subjects with Wilson disease or other Copper-related disorders.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-11-30 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 1 year
  Evaluated using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE)
Neutrophil Engraftment | 100 days
  Evaluate the time to neutrophil engraftment, defined as the first day in which absolute neutrophil count (ANC) >500/mm3 for three consecutive days
Overall Survival at Day 100, 6 months, and 1 year | Day 100, 6 months, and 1 year post-transplant
  Evaluate survival of subjects alive, with or without presence of disease, at the designated time points
Disease-Free Survival at Day 100, 6 months, and 1 year | Day 100, 6 months, and 1 year post-transplant
  Evaluate survival of subjects alive without disease at the designated time points

SECONDARY OUTCOMES:
Non-Relapse Mortality | Day 100
  Death that cannot be explained by persistence, relapse, or progression of underlying disease
Relapse Rate | Day 100, 6 months, 1 year
  Time to first relapse or progression of underlying disease after initiation of protocol therapy

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Mayer, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States